CLINICAL TRIAL: NCT01344174
Title: A Randomized, Open Label Study Evaluating the Efficacy and Safety of Glucocorticoids in Patients With Pre-ACLF-HBV
Brief Title: A Study Evaluating the Efficacy of Glucocorticoids in Patients With Pre-ACLF-HBV
Acronym: preACLF
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Third Military Medical University (Other)
Responsible Party: Xuqing Zhang, Department of infectious diseases, Southwest Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: preACLF2011
Record Dates: First submitted 2011-04-21; First posted 2011-04-28 (Estimated); Last update posted 2011-06-03 (Estimated); Status verified 2011-06

CONDITIONS: Liver Failure; Hepatitis B
Keywords: Acute-on-chronic liver failure; HBV; Dexamethasone; Prognosis
MeSH Terms: conditions — Liver Failure; Hepatitis B; Acute-On-Chronic Liver Failure | interventions — Lamivudine; Glutathione

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- glucocorticoids treatment (Other)
  Interventions: Drug: 5 days dexamethasone therapy

INTERVENTIONS:
Drug: 5 days dexamethasone therapy — dexamethasone 10mg, intravenously, po daily for the first 5 days
  Other Names: lamivudine; Transfusion of magnesium isoglycyrrhizinate injection; reduced glutathione; S-adenosyl-L- metionine

SUMMARY:
This is a randomized, open label study evaluating the efficacy and safety of glucocorticoids in patients with HBV associated pre-ACLF.

Sponsor: Department of infectious diseases, Southwest Hospital.

Indication: HBV associated acute-on-chronic pre-liver failure(pre-ACLF-HBV).

Objective: To evaluate the efficacy and safety of glucocorticoids in patients with pre-ACLF-HBV.

Trial Design: Randomized, open label study. Patients with pre-ACLF-HBV will be randomized 1:1 to One of the two groups:

A)Dexamethasone 10mg were intravenously injected po daily for the first 5 days, in combination with continued lamivudine 100mg po daily and traditional supporting treatments for 13 weeks. B)Control group. Any glucocorticoids will be not given in all patients. Continued lamivudine 100mg po daily and traditional supporting treatments will be given for 13 weeks.

Number of patients: Approximate number of patients to be randomized: N=200 (100 patients in each group).

Length of study: Screening period: 3 days; treatment period: 13 weeks.

Duration of study: 30 months after first patient randomized, including an recruitment period of 26 months.

Investigational treated regimen:Dexamethasone 10mg, iv, once day for 5 days.

Concomitant and Comparative regimen: Lamivudine 100mg po daily, traditional supporting treatments.

Assessments of Efficacy Primary endpoint: the survival rate at week 13. Secondary endpoint:①The levels of serum T-Bil ≤ 51.3µmol/L;②PTA >80%.

Safety: Adverse events, vital signs, and laboratory tests.

Procedures(summary): After signing informed consent and meeting screening parameters, patients will be randomized to one of the two treatment groups as described under trial design above. After randomization patients will be seen for evaluation at days 5,10,14,21,28,42,56,70,84,91.

Statistical analysis: Assume 1:1 randomization. The sample size is calculated for the primary efficacy variable, the survival rate. Assuming the survival rate equals to: 90% for group A and 50% for group B. 100 patients in each group are required to yield a 80% chance of detecting such a difference when a two-tailed test is employed at the 0.05 significance levels. Every eligible subject will be assigned with a randomization code and receive one of the two treatments, according to the sequence of enrolled.

DETAILED DESCRIPTION:
Synopsis of Protocol

Protocol of number: preACLF2011 Title: A randomized, open label study evaluating the efficacy and safety of glucocorticoids in patients with HBV associated pre-ACLF.

Sponsor: Department of infectious diseases, Southwest Hospital.

Indication: HBV associated acute-on-chronic pre-liver failure(pre-ACLF-HBV).

Objective: To evaluate the efficacy and safety of glucocorticoids in patients with pre-ACLF-HBV.

Trial Design: Randomized, open label study. Patients with pre-ACLF-HBV will be randomized 1:1 to one of the two groups: A)10mg dexamethasone were intravenously injected po daily for the first 5 days, in combination with continued lamivudine 100mg po daily and traditional supporting treatments for 13 weeks. B)Any glucocorticoids will be not given in all patients. Continued lamivudine 100mg po daily and traditional supporting treatments will be given for 13 weeks.

Number of patients: Approximate number of patients to be randomized: N=200 (100 patients in each group)

Length of study: Screening period: 3 days; treatment period: 13 weeks.

Duration of study: 30 months after first patient randomized, including an recruitment period of 26 months.

Investigational treated regimen: Short-term glucocorticoids treatment (10mg dexamethasone, iv, once day for the first 5 days).

Concomitant and comparative regimen treatments: Lamivudine 100mg po daily, traditional supporting treatments including: ①Transfusion of magnesium glycyrrhizinate injection (200mg, 1/d) and reduced glutathione (1200mg, 1/d); ②S-adenosyl-L- methionine (500 mg, intravenously, 2/d); ③Transfusion of human albumin (10 g, twice a week) and fresh frozen plasma (200 ml, twice a week); ④Nutritional supplements and prophylactic therapies for various complications being given.

Assessments of efficacy: Primary endpoint: the survival rate at week 13. Secondary endpoint: ①The levels of serum T-Bil ≤51.3µmol/L; ②PTA >80%.

Safety:Adverse events, vital signs, and laboratory tests.

Procedures(summary): After signing informed consent and meeting screening parameters, patients will be randomized to one of the two treatment groups as described under trial design above. After randomization patients will be seen for evaluation at days 5,10,14,21,28,42,56,70,84,91.

Statistical analysis Assume 1:1 randomization. The sample size is calculated for the primary efficacy variable, the survival rate. Assuming the survival rate equals to: 90% for group A and 50% for group B. 100 patients in each group are required to yield a 80% chance of detecting such a difference when a two-tailed test is employed at the 0.05 significance levels. Every eligible subject will be assigned with a randomization code and receive one of the two treatments, according to the sequence of enrolled.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients ≥18 and ≤ 65 years of age;
* serum hepatitis B surface antigen (HBsAg) being positive for at least 12 months;
* serum HBV DNA ≥104copies/ml, and did not receive any antiviral treatment with interferon or NA within 12 months;
* serum T-Bil≥171µmol/L;
* PTA>40%;
* serum ALT≥10×ULN in two weeks and >5×ULN at the initiation of treatment.

Exclusion Criteria:

* superinfection or coinfection with HAV, HCV, HDV,HEV, CMV, HIV, EBV;
* other liver diseases such as alcoholic liver disease, drug-induced hepatitis, Wilson disease, and autoimmune hepatitis;
* ascites determined by abdominal ultrasound scan;
* gastrointestinal bleeding or peptic ulcer or oesophageal varix;
* cirrhosis by abdominal ultrasound scan;
* bacterial or fungal infections;
* the malignant jaundice induced by obstructive or hemolytic jaundice;
* a history of diabetes or cardiac disease or hypertension or nephrosis.
* Inability or unwillingness to provide informed consent or abide the the requirements of the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2011-05; Primary Completion 2011-08 (Estimated); Study Completion 2013-11 (Estimated)

PRIMARY OUTCOMES:
Evidence of improving the survival rate of pre-ACLF-HBV by short-term glucocorticoids therapy | within 13 weeks after treatment

SECONDARY OUTCOMES:
Evidence of improving liver function of pre-ACLF-HBV | within 4 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Xuqing Zhang, Prof., Principal Investigator — Southwest Hospital, Third Military Medical University of China
Locations (1):
- Department of infectious disease, Southwest Hospital, Third Military Medical University, Chongqing, Chongqing Municipality, China